CLINICAL TRIAL: NCT02098668
Title: Model Driven Computation for Infertility Related Endocrinological Diseases - PAEON
Brief Title: Mathematical Model for the Human Menstrual Cycle, Endocrinological Diseases and Fertility Treatment-PAEON
Acronym: PAEON
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 17721_PAEON
Record Dates: First submitted 2013-06-18; First posted 2014-03-28 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Polycystic Ovary Syndrome; Endometriosis; Hyperprolactinemia
Keywords: menstrual cycle dynamics; PCOS; hyperprolactinemia; endometriosis; infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Endometriosis; Hyperprolactinemia; Infertility

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Probes to determine hormonal parameters
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Normal, pathological cycle, infertility: healthy women PCOS Endometriosis hyperprolactinemia fertility treatment
  Interventions: Other: Fertility treatment

INTERVENTIONS:
Other: Fertility treatment — Fertility treatment

SUMMARY:
Development of a bio-mathematical model of the human female cycle

DETAILED DESCRIPTION:
From hormonal measurements throughout 1-2 menstrual cycles in women with and without endocrinological pathology a mathematical model of the human menstrual cycle will be generated. The model will serve to predict development of the cycle including ovulation as well as to better understand the pathophysiology of endocrinological disorder. In a second step current treatment protocols for fertility treatment will be integrated into the model in order to optimize treatment outcome.

ELIGIBILITY:
Inclusion criteria:

- Women during their reproductive phase, no hormonal therapy

Exclusion criteria:

- Amenorrhoae

Ages: 18 Months to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women with normal and distrubed menstrual cycles Women receiving fertility treatment
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Hormonal parameters | 3 years
  Development of a mathematical model of the menstrual cycle

SECONDARY OUTCOMES:
Dynamics of fertility treatment | 2 years
  Mathematical model to improve fertility treatments

OTHER OUTCOMES:
Dynamics of gyneco-endocrinological diseases | 3 years
  To better understand the pathophysiological mechanisms in endocrinological diseases

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Leeners, MD, Principal Investigator — University Hospital Zurich, Division of Reproductive Endocrinology
Locations (1):
- University Hospital Zurich, Division of Reproductive Endocrinology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leeners B, Kruger THC, Geraedts K, Tronci E, Mancini T, Egli M, Roblitz S, Saleh L, Spanaus K, Schippert C, Zhang Y, Ille F. Associations Between Natural Physiological and Supraphysiological Estradiol Levels and Stress Perception. Front Psychol. 2019 Jun 11;10:1296. doi: 10.3389/fpsyg.2019.01296. eCollection 2019. PMID 31244718